CLINICAL TRIAL: NCT06881355
Title: Effect of Bruxism on the Clinical Success of Posterior Composite Restorations in Endodontically Treated Teeth: A Cross-sectional, Case-Control Study
Brief Title: Effect of Bruxism on the Clinical Success of Posterior Composite Restorations
Acronym: Bruxism
Status: Completed | Type: Observational
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Fatma Yilmaz, Asistant Professor Doctor, Muğla Sıtkı Koçman University
Other Study IDs: Brux-comp-1; MSKU-Resto-Brux-comp-1 (Other: MSKU)
Record Dates: First submitted 2025-03-04; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Bruxism; Wear, Occlusal; Fracture
Keywords: Bruxism; Posterior composite restoration; Clinical success; Endodontically tretaed tooth
MeSH Terms: conditions — Bruxism; Tooth Attrition; Fractures, Bone | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group-Bruxists with PCR post-ETT: Participants having previously undergone endodontic treatment and composite restorations on any of their posterior teeth and bruxism were assigned to the case group. The presence of bruxism was determined based on the participant's self-reported statements and intraoral findings.
  Interventions: Diagnostic Test: Bruxism diagnosis; Diagnostic Test: Clinical evaluation
- Control group-Non-bruxists with PCR post-ETT: Participants without bruxism and with PCR post-ETT were assigned to the control group.
  Interventions: Diagnostic Test: Bruxism diagnosis; Diagnostic Test: Clinical evaluation

INTERVENTIONS:
Diagnostic Test: Bruxism diagnosis — The presence of bruxism was determined based on the participant's self-reported statements and intraoral findings.
Diagnostic Test: Clinical evaluation — The PCRs on the relevant teeth were evaluated according to the revised FDI criteria

SUMMARY:
The goal of this study is to determine the effect of bruxism on the success of posterior composite restorations (PCRs) in endodontically treated teeth (ETT). The null hypotheses of present study were as follows: (1) bruxism would not have a significant effect on the success rate of PCRs in ETT; (2) other demographic and clinical variations, such as frequency of coloring agent usage, smoking habits, presence of pulpal pathology, periapical lesion, periodontal condition, antagonist tooth condition, cavity margin level, quality of endodontic treatment, enamel cracks, temporomandibular joint (TMJ) disorders, lateral occlusion scheme, institution where the restoration was performed, number of restored surfaces, and follow-up period, would not have a significant effect on the success rate of PCRs in ETT; and (3) functional, esthetic, and biological clinical success of PCRs of bruxists would not differ from that of non-bruxists. This cross-sectional, case-control study included 40 case patients (bruxists with PCR post-ETT) and 40 controls (non-bruxists). Sociodemographic characteristics and clinical findings were recorded. The PCRs on the relevant teeth were evaluated according to the revised FDI criteria.

DETAILED DESCRIPTION:
In studies that have conducted long-term follow-ups of posterior composite restorations (PCRs), the most common causes of failure are secondary caries, wear, and fractures. The success of PCRs is influenced by several factors: oral hygiene habits, caries risk, size of the carious lesion, occlusal relationships, presence of parafunctional habits, physical properties of the material used, tooth region in which the restoration is placed, size and location of the restoration, and chewing habits and forces. In addition, the literature suggests that PCRs have a low wear resistance. While this characteristic is considered to offer an advantage in the presence of parafunctional habits, its effect on the success of PCRs under excessive occlusal stress remains a subject of debate. There are many prospective and retrospective studies evaluating the performance of restorations; however, literature on the success of composite resin materials when applied as direct restorations of ETT in patients with bruxism is limited. Furthermore, with the continuous development and introduction of new adhesive techniques and improvements in the composition of composite resin materials, clinical studies need to be updated regularly to assess the performance of restorations.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-40 years, PCRs after endodontic treatment,
* Restorations up to 5 years,
* Class 1 and 2 restorations with a maximum of 3 wall loss according to cavity classification and not involving the cusps,
* Patients with low and moderate caries risk, and those with an occlusion classified as Class 1 Angle.

Exclusion Criteria:

* Teeth without antagonists;
* patients with crossbite; mobile teeth;
* teeth diagnosed with acute apical/periodontal abscess;
* presence of severe periodontal disease;
* presence of systemic diseases;
* pregnant and breastfeeding women;
* patients who had amalgam, post, or indirect methods chosen for definitive restoration after endodontic treatment;
* restorations performed more than 5 years ago;
* patients aged <18 or >40 years;
* restorations involving the cusps,
* patients with high caries risk, and non-dental plaque biofilm-induced gingival diseases.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: In this study, the initial data pool consists of patients who had undergone their first examination and had the necessary radiographs taken routinely. After clinically and radiographically identifying those who had underwent root canal treatment and composite restorations, the eligible participants were included in the study to evaluate their restorations.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Rate of Clinical success | 1-5 years-follow up period
  FDI scoring system

SECONDARY OUTCOMES:
% of patients with risk factors | 1-5 years-follow up period
  Clinical failure parameter

CONTACTS AND LOCATIONS:
Locations (1):
- Muğla Sıtkı Koçman University, Menteşe, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
sociodemographic characteristics and clinical findings
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Hickel R, Mesinger S, Opdam N, Loomans B, Frankenberger R, Cadenaro M, Burgess J, Peschke A, Heintze SD, Kuhnisch J. Revised FDI criteria for evaluating direct and indirect dental restorations-recommendations for its clinical use, interpretation, and reporting. Clin Oral Investig. 2023 Jun;27(6):2573-2592. doi: 10.1007/s00784-022-04814-1. Epub 2022 Dec 12. PMID 36504246
- [Background] van de Sande FH, Opdam NJ, Rodolpho PA, Correa MB, Demarco FF, Cenci MS. Patient risk factors' influence on survival of posterior composites. J Dent Res. 2013 Jul;92(7 Suppl):78S-83S. doi: 10.1177/0022034513484337. Epub 2013 May 20. PMID 23690354
- [Background] Manfredini D, Winocur E, Guarda-Nardini L, Paesani D, Lobbezoo F. Epidemiology of bruxism in adults: a systematic review of the literature. J Orofac Pain. 2013 Spring;27(2):99-110. doi: 10.11607/jop.921. PMID 23630682
- [Background] R.R. Moraes, M.S. Cenci, J.R. Moura, F.F. Demarco, B. Loomans, N. Opdam, Clinical performance of resin composite restorations, Curr. Oral Health Rep.9 (2022) 22-31.
- [Background] Hickel R, Manhart J. Longevity of restorations in posterior teeth and reasons for failure. J Adhes Dent. 2001 Spring;3(1):45-64. PMID 11317384
- [Background] Laske M, Opdam NJM, Bronkhorst EM, Braspenning JCC, Huysmans MCDNJM. Risk Factors for Dental Restoration Survival: A Practice-Based Study. J Dent Res. 2019 Apr;98(4):414-422. doi: 10.1177/0022034519827566. Epub 2019 Feb 20. PMID 30786222
- [Background] Kramer N, Reinelt C, Frankenberger R. Ten-year Clinical Performance of Posterior Resin Composite Restorations. J Adhes Dent. 2015 Aug;17(5):433-41. doi: 10.3290/j.jad.a35010. PMID 26525008
- [Background] Koyano K, Tsukiyama Y, Ichiki R, Kuwata T. Assessment of bruxism in the clinic. J Oral Rehabil. 2008 Jul;35(7):495-508. doi: 10.1111/j.1365-2842.2008.01880.x. PMID 18557916
- [Derived] Yilmaz F, Dorterler OC. Effect of Bruxism on the Clinical Success of Posterior Composite Restorations in Endodontically Treated Teeth: A Cross-Sectional, Case-Control Study. J Esthet Restor Dent. 2025 Oct;37(10):2180-2192. doi: 10.1111/jerd.70008. Epub 2025 Jul 27. PMID 40717393